CLINICAL TRIAL: NCT00633360
Title: The Oral Contraceptive Pill for Premenstrual Worsening of Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Hadine Joffe, MD, Vice Chair for Research, Psychiatry Department, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-P-002057
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Premenstrual Syndrome; Depression
Keywords: Women; PMS; Depression
MeSH Terms: conditions — Premenstrual Syndrome; Depression | interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drospirenone and ethinyl estradiol (Experimental)
  Interventions: Drug: Drospirenone and ethinyl estradiol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drospirenone and ethinyl estradiol — Once daily by mouth
  Other Names: Yaz
  Arms: Drospirenone and ethinyl estradiol
Drug: Placebo — Once daily by mouth
  Arms: Placebo

SUMMARY:
To determine if augmentation with the oral-contraceptive pill containing drospirenone and ethinyl estradiol is more effective than placebo in the treatment of premenstrual breakthrough of depression.

ELIGIBILITY:
Inclusion criteria

1. Women who are non-smokers between the ages of 18-45 years (smokers 18-34 years);
2. Regular menstrual cycles (26-34 days in length, predictable within 7 days) for the past 6 months;
3. Determination that the antidepressant medication was initiated for the treatment of unipolar major depression, minor depression (depression, not otherwise specified), or dysthymia. Major depression and dysthymia will be evaluated through administration of the Mini-International Neuropsychiatric Interview (MINI). Minor depression will be evaluated by administration of the Structured Clinical Interview for Diagnosis-IV(SCID)10 section J.3.
4. Use of an antidepressant for at least 3 months for treatment of a depressive disorder, with stable dose for at least 2 months. It is acceptable to be on more than one psychiatric medication as long as one of them is an antidepressant.
5. Expected continued use of the same antidepressant at the same dose for the duration of the study;
6. 30% increase of the mid-follicular phase Montgomery-Åsberg Depression Rating Scale (MADRS) score to the late-luteal phase MADRS will be required for eligibility during the tracking phase of the study and will be assessed prospectively over 1 menstrual cycle.
7. Normal pelvic exam and PAP smear in the past 12 months;
8. Normal TSH at screen - if on thyroid medication, must be on a stable dose for 2 months or greater, and have a normal TSH at screen;
9. Negative serum HCG at baseline, and negative urine HCG at visits 3 and 5;
10. Normal potassium (K) levels at screen;
11. Willingness to use barrier contraceptive methods during the study, if sexually active;
12. Good general health.

Exclusion Criteria:

1. Amenorrhea or irregular menstrual periods (defined as unable to predict within 7 days) during past 6 months
2. Pregnancy or breastfeeding (serum HCG test administered at baseline study visit, and urine HCG at visits 3 and 5)
3. Current cigarette smoking in women who are older than 34 years
4. Presence of any of the following psychiatric and substance use disorders, based on administration of the MINI at the baseline study visit:

   Any history of mania or hypomania suggesting bipolar disorder Any lifetime history of a psychotic disorder
5. Depression deemed by the physician investigator to be too severe to be treated in the study
6. Use of benzodiazepines or antipsychotic to target premenstrual symptoms
7. Luteal-phase dose adjustment of the antidepressant. Use of a hormone releasing IUD (intrauterine device)
8. Use of an OCP or other systemic hormonal therapies (oral, transdermal or injection preparations of androgens, estrogens, or progestins) in the past 2 months;
9. Any contraindication or previous adverse event to any OCP therapy;
10. Current use of ketoconazole, rifampin, carbamazepine, topiramate, oxcarbazepine, modafinil, phenytoin, or phenobarbital (because of interaction with hormonal therapy).
11. Current use of potassium-sparing agents, such as potassium-sparing diuretics (e.g., spironolactone), ACE inhibitors, angiotensin-II receptor antagonists, heparin, aldosterone antagonists, NSAIDS, potassium sparing diuretics or potassium-supplements (because of risk of developing arrhythmia with two potassium-elevating agents).
12. Hepatic dysfunction, renal insufficiency, pulmonary, adrenal, or metabolic diseases (including elevated serum potassium levels, if known) that may put subject at risk when treated with study medication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadine Joffe, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Drospirenone and Ethinyl Estradiol: Drospirenone and ethinyl estradiol
  Drospirenone and ethinyl estradiol: Once daily by mouth
- Placebo: Placebo
  Placebo: Once daily by mouth
Period: Overall Study
Arm/Group | Drospirenone and Ethinyl Estradiol | Placebo
Started | 16 | 16
Completed | 12 | 13
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drospirenone and Ethinyl Estradiol | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (7.3) | 26.3 (7.1) | 27.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Luteal Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Åsberg Depression Rating Scale is a widely used 10-item clinician-rated scale that describes the severity of depressive symptoms. It has a range of 0-60 with higher scores indicating greater symptom burden. Participants were assessed at baseline and during 2nd treatment month in order to calculate the change in MADRS score.
Time Frame: Baseline and 2 months
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Drospirenone and Ethinyl Estradiol | Placebo
Number analyzed (Participants) | 12 | 13
percent change | -43.6 [-73.8 to -24.6] | -38.9 [-61.5 to 0.0]
Statistical Analysis 1: Comparison: Drospirenone and Ethinyl Estradiol vs Placebo; Test type: Superiority or Other; p = .59, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent Change in Daily Record of Severity of Problems (DRSP)
Description: The DRSP is a 24-item self-administered daily dairy that assesses the severity of mood and physical symptoms which occur as part of the premenstrual syndrome and PMDD. Each question is rated on a scale of 1-6 with a total score range from 24-144. A higher score indicates greater symptom burden.
Time Frame: Baseline and 2 months
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Drospirenone and Ethinyl Estradiol: Drospirenone and ethinyl estradiol
- Placebo: Placebo
Arm/Group | Drospirenone and Ethinyl Estradiol | Placebo
Number analyzed (Participants) | 12 | 13
percent change | -23.5 [-38.4 to -7.0] | -20.9 [-38.7 to -11.7]
Statistical Analysis 1: Comparison: Drospirenone and Ethinyl Estradiol vs Placebo; Test type: Superiority or Other; p = .29, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Drospirenone and Ethinyl Estradiol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 10/16 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drospirenone and Ethinyl Estradiol (N=16) | Placebo (N=16)
spotting (Reproductive system and breast disorders) | 8 (8) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
headache (Nervous system disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No